CLINICAL TRIAL: NCT00006173
Title: Assessment of Renal Artery Stenosis and Renovascular Hypertension by Contrast Enhanced Magnetic Resonance Imaging: A Pilot Study
Brief Title: Magnetic Resonance Imaging for Evaluating Kidney Function
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000195; 00-CC-0195
Record Dates: First submitted 2000-08-11; First posted 2000-08-14 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-01

CONDITIONS: Healthy; Renovascular Hypertension
Keywords: Atherosclerosis; Hypertension; Magnetic Resonance Angiography
MeSH Terms: conditions — Hypertension, Renovascular; Atherosclerosis; Hypertension

SUMMARY:
Renovascular hypertension (RVH) is a potentially curable disease affecting 0.5-5 percent of patients with hypertension. The current diagnostic work-up of RVH involves a complex algorithm which includes doppler ultrasound, captopril renography and conventional angiography. Because of the expense, risk and inconvenience of this workup, patients may not be correctly diagnosed.

Advances in MR technology present the opportunity to develop a single comprehensive test. This would combine an MR angiogram that provides anatomic information about the renal arteries, and an MR renogram that provides information about the functional impact of a stenosis as a cause of hypertension. Our main purpose is to test MR renography with and without an oral angiotensin converting enzyme inhibitor (ACEI) combined with MR angiography against the reference standard of captopril radionuclide renography. Secondary goals of this study are to test whether hypoxia within ischemic kidneys affected by RVH is detectable by T2 weighted (Blood oxygen level dependent or BOLD) MRI. This is considered of value since such a test of oxygenation would further shorten and simplify the diagnostic MR test. Information gained from this study could lead to important changes in the diagnostic and pathophysiologic understanding of RVH.

DETAILED DESCRIPTION:
Renovascular hypertension (RVH) is a potentially curable disease affecting 0.5-5% of patients with hypertension. The current diagnostic work-up of RVH involves a complex algorithm which includes doppler ultrasound, captopril renography and conventional angiography. Because of the expense, risk and inconvenience of this workup, patients may not be correctly diagnosed.

Advances in MR technology present the opportunity to develop a single comprehensive test. This would combine an MR angiogram that provides anatomic information about the renal arteries, and an MR renogram that provides information about the functional impact of a stenosis as a cause of hypertension. Our main purpose is to test MR renography with and without an oral angiotensin converting enzyme inhibitor (ACEI) combined with MR angiography against the reference standard of captopril radionuclide renography. Secondary goals of this study are to test whether hypoxia within ischemic kidneys affected by RVH is detectable by T2* weighted (Blood oxygen level dependent or BOLD) MRI. This is considered of value since such a test of oxygenation would further shorten and simplify the diagnostic MR test. Information gained from this study could lead to important changes in the diagnosis and pathophysiologic understanding of RVH.

ELIGIBILITY:
INCLUSION CRITERIA

Healthy volunteers or patients with significant clinical suspicion of renovascular hypertension.

Subjects able to understand the informed consent for this study.

Subjects must be able to hold their breath for 20 second intervals.

Patients must be clinically stable and be judged by their physician able to tolerate the MR study of 1.5-2 hour duration.

EXCLUSION CRITERIA

Any contraindication for MR study including: pacemaker or other implanted electronic device; cochlear implants; metal in the eye; embedded shrapnel fragments; cerebral aneurysm clips; or medical infusion pumps.

Allergy to gadolinium, iodinated contrast media, ACEIs, or sulphur-containing medication.

Patients have a hematocrit at or below 30. Severe anemia may predispose to hypotension after captopril.

Patients with hyperkalemia (plasma potassium: above 5.0 mmol/L), because of the risk of arrhythmia.

Clinically unstable patients and those unable to tolerate a 1-2 hour MR study. Examples of medical conditions that would lead to exclusion include unstable angina, dyspnea at rest, severe pain at rest, or severe back pain.

Pregnancy.

Nursing mothers.

Subjects who are claustrophobic and are unable to tolerate MR imaging.

Patients with a serum creatinine concentration above 4mg/dl.

Bilateral renal stents.

Healthy subjects must not have an abnormality detected on dipstick urinalysis, or a systolic BP above 140 mmHg or a diastolic BP above 90 mmHg on screening examination or an abnormal BUN or creatinine level in the blood.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2000-08; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kulkarni S, O'Farrell I, Erasi M, Kochar MS. Stress and hypertension. WMJ. 1998 Dec;97(11):34-8. PMID 9894438
- [Background] Bouyounes BT, Libertino JA. Renovascular hypertension. Curr Opin Urol. 1999 Mar;9(2):111-4. doi: 10.1097/00042307-199903000-00004. PMID 10726080
- [Background] Taylor A. Radionuclide renography: a personal approach. Semin Nucl Med. 1999 Apr;29(2):102-27. doi: 10.1016/s0001-2998(99)80003-8. PMID 10321824